CLINICAL TRIAL: NCT01467557
Title: 1•DAY ACUVUE® TruEye™ Brand Contact Lenses & 1•DAY ACUVUE® MOIST® Brand Contact Lenses With LACREON® TECHNOLOGY Daily Disposable Performance Overview Registry -TEMPO Study
Brief Title: Daily Disposable Performance of 1•DAY ACUVUE® TruEye™ and 1•DAY ACUVUE® MOIST® With LACREON® TECHNOLOGY
Acronym: TEMPO
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-005059
Record Dates: First submitted 2011-10-26; First posted 2011-11-08 (Estimated); Results first posted 2015-09-15 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2015-10

CONDITIONS: Myopia; Hyperopia
Keywords: adverse events
MeSH Terms: conditions — Myopia; Hyperopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1-Day ACUVUE TruEye contact lens users: 1-Day ACUVUE TruEye contact lens users
  Interventions: Device: narafilcon B daily disposable soft contact lenses
- 1-Day ACUVUE MOIST contact lens users: 1-Day ACUVUE MOIST contact lens users
  Interventions: Device: etafilcon A daily disposable soft contact lenses

INTERVENTIONS:
Device: narafilcon B daily disposable soft contact lenses — daily disposable soft contact lenses
  Other Names: 1-Day ACUVUE TruEye
  Groups: 1-Day ACUVUE TruEye contact lens users
Device: etafilcon A daily disposable soft contact lenses — daily disposable soft contact lenses
  Other Names: 1-Day ACUVUE MOIST
  Groups: 1-Day ACUVUE MOIST contact lens users

SUMMARY:
This study is an observational registry of patients who have recently been prescribed 1•DAY ACUVUE® TruEye® or 1•DAY ACUVUE® MOIST® Brand Contact Lenses with LACREON® TECHNOLOGY.

ELIGIBILITY:
Inclusion Criteria:

* Wearers of 1•DAY ACUVUE® TruEye™ or 1•DAY ACUVUE® MOIST® daily disposable soft contact lenses in both eyes aged >8 years of age who have recently begun use of that lens type and have purchased at least 3 month supply of lenses.
* The registrant must read and sign the Informed Consent form. Minor subjects must obtain parental signature of Informed Consent and also sign an Informed Assent Form.
* The registrant must sign the Release of Medical Records in the event of an adverse event in the study.
* The registrant must appear able and willing to adhere to the instructions set forth in this clinical protocol.

Exclusion Criteria:

* Previously wearing the type of lenses with which they are registering (1•DAY ACUVUE® TruEye™ or 1•DAY ACUVUE® MOIST® Daily Disposable lenses).
* Current participant in an unrelated research study.
* Employee or family member of Recruiting Practitioner or Johnson & Johnson.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have recently been fit with 1-Day ACUVUE® TruEye™ or 1- Day ACUVUE® MOIST® daily disposable lenses.
Sampling Method: Non-Probability Sample
Enrollment: 1171 (Actual)
Dates: Start 2011-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - Campbell, California
  - Fullerton, California
  - Huntington Beach, California
  - Los Angeles, California
  - Mountain View, California
  - Newport Beach, California
  - Salinas, California
  - San Francisco, California
  - San Jose, California
  - Sunnyvale, California
  - Washington D.C., District of Columbia
  - Boca Raton, Florida
  - Fort Lauderdale, Florida
  - North Miami, Florida
  - Pembroke Pines, Florida
  - Wellington, Florida
  - Roswell, Georgia
  - Des Moines, Iowa
  - Shreveport, Louisiana
  - Belmont, Massachusetts
  - Cambridge, Massachusetts
  - Dedham, Massachusetts
  - Lake Hopatcong, New Jersey
  - New York, New York
  - Charlotte, North Carolina
  - Gastonia, North Carolina
  - Cleveland, Ohio
  - Johnstown, Ohio
  - Westerville, Ohio
  - Brentwood, Tennessee
  - Amarillo, Texas
  - Milwaukee, Wisconsin

REFERENCES:
- [Derived] Hickson-Curran SB, Chalmers RL, Keay L, Gleason W. Patient-Reported Wearing Experience From Hydrogel Daily Disposable Wearers Older Than 40 Years From the TEMPO Registry. Eye Contact Lens. 2017 Sep;43(5):313-317. doi: 10.1097/ICL.0000000000000271. PMID 27243356
- [Derived] Chalmers RL, Hickson-Curran SB, Keay L, Gleason WJ, Albright R. Rates of adverse events with hydrogel and silicone hydrogel daily disposable lenses in a large postmarket surveillance registry: the TEMPO Registry. Invest Ophthalmol Vis Sci. 2015 Jan 8;56(1):654-63. doi: 10.1167/iovs.14-15582. PMID 25574042

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1-Day ACUVUE TruEye Contact Lens Users | 1-Day ACUVUE MOIST Contact Lens Users
Started | 601 | 570
2 Week Survey Completed | 551 | 522
4 Month Survey Completed | 533 | 493
12 Month Survey Completed | 502 | 463
Completed | 502 | 463
Not Completed | 99 | 107

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1-Day ACUVUE TruEye Contact Lens Users | 1-Day ACUVUE MOIST Contact Lens Users | Total
Number analyzed (Participants) | 601 | 570 | 1171
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 106 | 121 | 227
  Between 18 and 65 years | 484 | 445 | 929
  >=65 years | 11 | 4 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (13.9) | 30.3 (12.9) | 31.8 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 400 | 392 | 792
  Male | 201 | 178 | 379
Region of Enrollment [Number; unit: participants]
  United States | 601 | 570 | 1171

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Description: Adverse events were reported by subjects via the electronic surveys if they responded "yes" to the question "Since we last contacted you, have you experienced a red or painful eye that required a visit to an eye doctor or emergency room?". Consensus diagnosis was made after review of clinical records by Adjudication Panel.
Time Frame: Self-report at 2 Week, 4 Month or 12 Month surveys
Population: The analysis population consisted of subjects that were enrolled into this study. (i.e subjects that met all study eligibility criteria)
Measure: Number; unit: participants
Groups:
- 1-Day ACUVUE TruEye Contact Lens Users: 1-Day ACUVUE TruEye contact lens users
  narafilcon B daily disposable soft contact lenses: daily disposable soft contact lenses.
  Registered Wearers who had been recently fit with these daily disposable lenses.
- 1-Day ACUVUE MOIST Contact Lens Users: 1-Day ACUVUE MOIST contact lens users
  etafilcon A daily disposable soft contact lenses: daily disposable soft contact lenses.
  Registered Wearers who had been recently fit with these daily disposable lenses.
Arm/Group | 1-Day ACUVUE TruEye Contact Lens Users | 1-Day ACUVUE MOIST Contact Lens Users
Number analyzed (Participants) | 601 | 570
participants
  Corneal Infiltrative Events | 2 | 0
  CL-Related Adverse Events with Office Visit | 8 | 3
  Not CL-Related Adverse Events with Office Visit | 5 | 2
  "Yes" to Red Eye Question, but no Office Visit | 6 | 5

2. Secondary Outcome: Change in 8-item Contact Lens Dry Eye Questionnaire Score From Baseline to 2 Week, 4 Month and 12 Month Surveys
Description: The response set for each question was a 5-level likert scale. Intensity of discomfort, dryness, blurriness were measured with the likert scale from 0(Never Have It) to 5(Very Intense). Frequency of discomfort, dryness, blurry vision, removal of lenses, and eye closure(how often you wanted to close them) were measured with the likert scale from 1(Never) to 5(Constantly). The sum of all responses was recorded for each subject and then the average sum for all subjects was reported. The average can range from 0- 40 (continuous).
Time Frame: Baseline, 2 Week, 4 Month or 12 Month surveys
Population: The analysis population consists of all subjects that were considered to be experienced contact lens wearers. Subjects were considered to be experienced contact lens wearers if subjects were assigned daily disposable lens at all evaluation points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1-Day ACUVUE TruEye Contact Lens Users | 1-Day ACUVUE MOIST Contact Lens Users
Number analyzed (Participants) | 418 | 400
units on a scale
  Baseline, n=368, 320 | 12.8 (7.2) | 12.3 (7.2)
  2 weeks, n=418,400 | 7.3 (5.2) | 8.0 (5.5)
  4 months, n=418,400 | 8.7 (5.7) | 9.3 (6.2)
  12 months, n=418,400 | 9.0 (6.3) | 9.2 (6.1)

ADVERSE EVENTS:
Arm/Group | 1-Day ACUVUE TruEye Contact Lens Users | 1-Day ACUVUE MOIST Contact Lens Users
Serious Adverse Events (participants affected / at risk) | 0/601 | 0/570
Other Adverse Events (participants affected / at risk) | 0/601 | 0/570

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days